CLINICAL TRIAL: NCT04498000
Title: Analysis of the Pachychoroid Phenotype in an Asian Population
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Gemmy Cheung Chui Ming, Professor, Singapore National Eye Centre
Other Study IDs: R1661/58/2019
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pachychoroid Disease
Keywords: pachychoroid neovasculopathy; pachychoroid choroidal vasculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The understanding of pachychoroid phenotype is incomplete. It is important to understand the risk of conversion from an uncomplicated pachychoroid phenotype to the pachychoroid disease phenotype, to guide appropriate management of these patients.

DETAILED DESCRIPTION:
The progression of uncomplicated pachychoroid phenotype to pachychoroid disease is not well established and the pathophysiology of these phenotypes remains unknown: specifically if the occurence of pachyvessels is the primary event, or develops secondary to the inner choroidal attenuation.

A longitudinal study of the pachychoroid phenotype will provide much needed information regarding the natural history of the pachychoroid phenotype. Secondly, a detailed chronicle of the choroidal alterations in the pachychoroid disease spectrum may yield insights into the pathogenesis, and facilitate the development of disease modulation strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of uncomplicated and/or non-neovascular pachychoroid phenotype in at least one eye.
2. Subfoveal choroidal thickness >300 microns on enhanced depth imaging optical coherence tomography for at least one eye
3. Male or female patients above 45 years of age
4. Willingness to undergo pupil dilation, and protocol- required procedures for both eyes
5. Willing to provide written informed consent

Exclusion Criteria:

1. Presence of disorders of the ocular media which interfere with visual acuity and other ocular assessments, including Spectral domain- optical coherence tomography during the study period
2. Pregnant or nursing women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit 120 participants from the Singapore National Eye Centre (SNEC) and National University Hospital (NUH). SNEC will recruit 70 participants and NUH will recruit 50 participants for this study. There is no subject restriction based on race of the subject.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of progression of pachychoroid phenotypes in 2 subtypes | 2 years observation
  Two subtypes of pachychoroid phenotypes:
  1. from an uncomplicated pachychoroid phenotype, to a pachychoroid disease entity
  2. from non neo-vascular pachychoroid disease, to neovascular pachychoroid disease
Risk factors for progression in 2 subtypes of pachychoroid phenotypes | 2 years
  1. from an uncomplicated pachychoroid phenotype, to a pachychoroidal disease entity
  2. from neo-vascular pachychoroid disease, to neovascular pachychoroid disease
Assess the chronology of choroidal changes in patients | 2 years
  Determine the occurence of pachyvessles is the primary event, or consequent to inner choroidal attenuation

CONTACTS AND LOCATIONS:
Overall Officials: Xinyi Su, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore National Eye Centre, Singapore

IPD SHARING:
Plan to Share IPD: No